CLINICAL TRIAL: NCT01447862
Title: Vernakalant Versus Ibutilide In Recent-Onset Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Hans Domanovits, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Verna-Ibu-AF
Record Dates: First submitted 2011-10-05; First posted 2011-10-06 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Atrial Fibrillation
Keywords: recent-onset
MeSH Terms: conditions — Atrial Fibrillation | interventions — vernakalant; ibutilide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vernakalant (Active Comparator): Initially, patients will be given 3mg/kg Vernakalant in 100ml normal saline over 10min. If atrial fibrillation continues after another 15 minutes of observation, patients will receive a second infusion of Vernakalant (2mg/kg), again over 10 minutes. If the initial rhythm has not converted to sinus rhythm after 2 hours, consented patients will be treated with electrical cardioversion using a standard routine protocol.
  Interventions: Drug: Brinavess (Vernakalant)
- Ibutilide (Active Comparator): Patients will be given 1mg of ibutilide in 100ml normal saline intravenously over 10min. If atrial fibrillation continues after another 10 minutes of observation, patients will receive a second infusion of 1mg ibutilide, again over 10min. If the initial rhythm has not converted to sinus rhythm after 2 hours, consented patients will be treated with electrical cardioversion using a standard routine protocol.
  Interventions: Drug: Corvert (Ibutilide)

INTERVENTIONS:
Drug: Brinavess (Vernakalant) — 3mg/kg Brinavess (Vernakalant) in 100ml normal saline over 10min. If atrial fibrillation continues after another 15 minutes of observation, patients will receive a second infusion of 2mg/kg Brinavess (Vernakalant) over 10 minutes
  Arms: Vernakalant
Drug: Corvert (Ibutilide) — Patients will be given 1mg of Corvert (Ibutilide) in 100ml normal saline intravenously over 10min. If atrial fibrillation continues after another 10 minutes of observation, patients will receive a second infusion of 1mg ibutilide over 10min.
  Arms: Ibutilide

SUMMARY:
Atrial fibrillation is the most common cardiac arrhythmia and is expected to affect about 30 million North Americans and Europeans by 2050. Atrial fibrillation is associated with increased cardiovascular morbidity and mortality, with stroke being an especially important and potentially devastating complication. Many studies have investigated the efficacy of different drugs in converting atrial fibrillation to sinus rhythm. There are numerous randomized controlled trials that have tested the efficacy of agents against placebo and some trials that directly compared the efficacy of two or more different drugs. The class III antiarrhythmic drug Ibutilde is approved for the acute termination of atrial fibrillation and atrial flutter of recent onset and has been shown to be superior to sotalol and equivalent to flecainide in this indication. Recently, the relatively atrial selective antiarrhythmic agent vernakalant has been approved by the European Commission for the rapid conversion of recent onset AF to sinus rhythm in adults. The investigators hypothesize that the period of time needed for cardioversion to sinus rhythm and the efficacy of cardioversion within 90 minutes is different between vernakalant and ibutilide in patients with recent-onset atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of atrial fibrillation since no longer than 48 hours
* Age 18 - 90 years

Exclusion Criteria:

* Need for immediate electrical cardioversion due to hemodynamic instability (hypotension: systolic blood pressure < 100 mmHg, dyspnea, loss of consciousness, unstable angina)
* Moderate to severe heart failure (NYHA III/IV) and patients with previously documented left ventricular ejection fraction (LVEF) ≤ 35%
* History or signs of acute coronary syndromes (acute myocardial infarction, unstable angina) within the last 30 days
* Resting ventricular rate < 80 beats per minute without pace maker back-up
* QT interval of > 440 milliseconds
* Wolff-Parkinson-White (WPW) syndrome
* History of Torsade de pointes arrhythmias or other polymorphic ventricular tachycardias
* Signs of thyreotoxicosis
* Sick Sinus Syndrome or atrioventricular block greater than first degree
* Severe valvular heart disease, clinically meaningful hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy, or constrictive pericarditis
* Serious disorders of the hepatic, renal (Creatinine > 2.5mg/dl), pulmonary, gastrointestinal, hematologic or central nervous system and serious psychiatric disorders
* Abnormal serum electrolytes despite adequate therapy (especially potassium <3.5 mmol/l or > 5.5 mmol/l)
* Intravenous use of other Class I or III antiarrythmic drugs within 4 hours of study drug application
* Pregnancy (a β-HCG test will be performed in all female subjects apart from women > 50 years and with amenorrhea for at least 12 month (absence of other causes of amenorrhoea)
* Known hypersensitivity to study medication

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Time in minutes until conversion to sinus rhythm (measured from the start of the first study drug administration) | 90 minutes

SECONDARY OUTCOMES:
Conversion rate to sinus rhythm within 90 minutes (measured from the start of the first study drug administration) | 90 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Emergency Medicine, Vienna, Vienna, Austria

REFERENCES:
- [Background] Camm AJ, Capucci A, Hohnloser SH, Torp-Pedersen C, Van Gelder IC, Mangal B, Beatch G; AVRO Investigators. A randomized active-controlled study comparing the efficacy and safety of vernakalant to amiodarone in recent-onset atrial fibrillation. J Am Coll Cardiol. 2011 Jan 18;57(3):313-21. doi: 10.1016/j.jacc.2010.07.046. PMID 21232669
- [Background] Domanovits H, Schillinger M, Thoennissen J, Nikfardjam M, Janata K, Brunner M, Laggner AN. Termination of recent-onset atrial fibrillation/flutter in the emergency department: a sequential approach with intravenous ibutilide and external electrical cardioversion. Resuscitation. 2000 Aug 1;45(3):181-7. doi: 10.1016/s0300-9572(00)00180-5. PMID 10959017
- [Background] Stiell IG, Dickinson G, Butterfield NN, Clement CM, Perry JJ, Vaillancourt C, Calder LA. Vernakalant hydrochloride: A novel atrial-selective agent for the cardioversion of recent-onset atrial fibrillation in the emergency department. Acad Emerg Med. 2010 Nov;17(11):1175-82. doi: 10.1111/j.1553-2712.2010.00915.x. PMID 21175515
- [Derived] Simon A, Niederdoeckl J, Skyllouriotis E, Schuetz N, Herkner H, Weiser C, Laggner AN, Domanovits H, Spiel AO. Vernakalant is superior to ibutilide for achieving sinus rhythm in patients with recent-onset atrial fibrillation: a randomized controlled trial at the emergency department. Europace. 2017 Feb 1;19(2):233-240. doi: 10.1093/europace/euw052. PMID 28175295